CLINICAL TRIAL: NCT00223665
Title: A Prospective Study of Intermittent Androgen Suppression (IAS) in Men With Localized Prostate Cancer Who Have Biochemical Relapse After Radiation Therapy or Radical Prostatectomy
Brief Title: Effects of IAS in Men With Localized Biochemical Relapsed Prostate Cancer
Acronym: IAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Celestia Higano, Professor, Medicine, Division of Oncology & Urology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30296; 973730AC06 (Other: University of Washington, HSRC Approval #); HSD 30296 (Other: University of Washington, Human Subjects IRB #)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: Intermittent Hormone Therapy; Intermittent Androgen Suppression; Biochemical Relapsed Prostate Cancer; Androgen Deprivation Therapy; Localized Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Intervention Model Description: All subjects underwent androgen suppression with a two-week lead-in of Flutamide, followed by 9 monthly injections of Leuprolide Acetate. If PSA reached the appropriate nadir at by month 9, the androgen suppression was interrupted. Once the PSA reached the appropriate threshold, the subjects resumed treatment for another 9 months. These cycle continued until the patient withdrew from the study, was taken off the study due to toxicities or the decision of the investigator, or until the treatment with IAS was no longer effective in controlling the prostate cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intermittent Androgen Suppression (IAS) (Experimental): Intermittent Androgen Suppression in 9 month cycles with a combination of a two-week lead-in of Flutamide, followed by 9 monthly injections of Leuprolide Acetate.
  Flutamide dosed as 250mg orally three times a day for 14 days prior to the initiation of Leuprolide Acetate.
  Leuprolide Acetate dosed as 7.5mg intramuscular (IM) injections once per month for a total of 9 months.
  Interventions: Drug: Flutamide; Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Flutamide — Flutamide dosed at 250mg orally three times a day for 14 days prior to the initiation of Leuprolide Acetate.
  Other Names: Eulexin
Drug: Leuprolide Acetate — Leuprolide Acetate dosed at 7.5mg intramuscular (IM) injections once per month for a total of 9 months.
  Other Names: Lupron Depot; Eligard; Lupron

SUMMARY:
This study was a prospective analysis in men with localized prostate cancer who had rising Prostate Specific Antigen (PSA) levels after definitive treatment with surgery or radiation. Patients received Intermittent Androgen Suppression (IAS) in 9 month cycles until they became metastatic, became castrate resistant, or withdrew from the study. Subjects were monitored for time to development of Castration Resistant Prostate Cancer (CRPC) and overall survival. They were also monitored for the impact of IAS on a variety of neuro-psychiatric assessments and on bone density.

DETAILED DESCRIPTION:
The standard first line treatment for men with early stage newly diagnosed localized prostate cancer is a surgical removal of the prostate, localized external beam radiation, brachytherapy, or a combination of surgery and radiation. In most patients Prostate Specific Antigen (PSA) levels will decline after these localized treatments, demonstrating a response to these therapies. However despite an initial response to localized treatment, some men will go on to later develop a rise in PSA levels, an indicator of Biochemical Relapsed Prostate Cancer (BRPC). For BRPC patients who have not yet developed metastasis, the standard treatment is Androgen Deprivation Therapy (ADT) to decrease levels of Testosterone, subsequently decreasing PSA levels. A low value for the PSA is more desirable as it may indicate no tumor growth.

ADT may be administered as a continuous treatment (Continuous Androgen Suppression, or CAS) or as intermittent treatment (Intermittent Androgen Suppression, or IAS). This treatment is continued until the development of Castration Resistant Prostate Cancer (CRPC), indicated by a rise in PSA despite ADT. Giving the hormone therapy intermittently (in cycles of treatment and off treatment periods) appears to delay the change of prostate cancer to a type of prostate cancer that resists hormone therapy, prolonging efficacy of ADT monotherapy. IAS may also decrease the impact of ADT on mental status.

This study evaluated the effect of intermittent androgen suppression on time to androgen independent progression (the development of castration resistant disease) and overall survival in men with localized prostate cancer. Subjects were also evaluated for the effects of intermittent androgen suppression on a variety of neuro-psychiatric assessments and on bone density.

The subjects in this study had a rising PSA value after definitive therapy either with radical prostatectomy or external beam irradiation for the treatment of prostate cancer. All subjects were males at or over the age of 21 years.

New subjects were introduced to this study protocol (along with other non-study treatment options) during a clinic visit with Dr. Higano or another sub-investigator. After informed consent was obtained, subjects underwent the following screening procedures before starting treatment: Bone density scan (DEXA), Technetium-99 bone scan, CT scan of the chest, abdomen, and pelvis, blood draw, and neuro-psychiatric assessments. Subjects then began androgen suppression with a two-week lead-in of Flutamide, followed by 9 monthly injections of Leuprolide Acetate. During the treatment, they had quarterly clinic visits and blood draws. Their PSA levels were monitored monthly, and if their PSA reached the appropriate nadir at by month 9, the androgen suppression was interrupted. At the end of each treatment cycle, subjects underwent another bone density test, blood draw, problem solving test, and neuro-psychiatric assessments.

During the "off treatment" phase, the subject will again had quarterly clinic visits, blood draws, and neuro-psychiatric assessments. PSA and testosterone were be monitored monthly. Once the PSA reached the appropriate threshold, the subject performed another set of screening procedures and resumed treatment for another 9 months. This cycle continued until the patient withdrew from the study, was taken off the study due to toxicities or the decision of the investigator, or until the treatment with IAS was no longer effective in controlling the prostate cancer. The neuro-psychiatric assessments were only performed during the subject's first cycle of treatment (consisting of the 9 months on treatment, and at month 3 of the off treatment period afterwards).

ELIGIBILITY:
Inclusion Criteria:

* Biochemical relapse (rising PSA) after initial treatment (radiation therapy, brachytherapy, or radical prostatectomy) for histologically or cytologically confirmed adenocarcinoma of the prostate
* Clinical stage A2, B, C, D1
* Age: older than 21 years old
* Performance status of 0 or 1
* Pretreatment serum testosterone, normal range (or no clinical evidence of testosterone deficiency).
* If less than 30 months since completion of radiation therapy, biopsy of prostate suggested within 6 months of study entry. If more than or equal to 30 months since completion of radiation therapy, biopsy of prostate suggested within 1 year.
* Written informed consent.

Exclusion Criteria:

* Abnormal bone scan suggestive of metastatic osseous disease.
* Previous hormonal manipulation including orchiectomy or any medication with significant antiandrogenic activity (combined androgen suppression over 9 months, monotherapy antiandrogens, estrogens, ketoconazole). *Neoadjuvant androgen suppression therapy of less than or equal to 3 months is allowed, if this androgen suppression therapy was completed more than or equal to 1 year prior to study enrollment AND if the Testosterone level is within the normal ranges.
* Any systemic chemotherapy or curative radiotherapy within 6 months.
* Hepatic dysfunction:

  * Total bilirubin greater than 2.0 mg/dl
  * Aspartate transaminase (AST; SGOT) greater than 3 times the upper limit of normal range
  * Lactate dehydrogenase (LDH) greater than 3 times the upper limit of normal range).
* Renal dysfunction:

  * Blood urea nitrogen (BUN) greater than 40 mg/dl
  * Serum Creatinine greater than 2.0 mg/dl.
* History or presence of other malignancy within the last 5 years (except treated squamous/basal cell carcinoma of the skin or superficial bladder carcinoma).
* Hypersensitivity to flutamide or leuprolide.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 1997-01-08 (Actual); Primary Completion 2012-09-06 (Actual); Study Completion 2012-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celestia Higano, MD, Principal Investigator — University of Washington
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo KF, Hunter-Merrill R, Gulati R, Hall SP, Gambol TE, Higano CS, Yu EY. Relationships between times to testosterone and prostate-specific antigen rises during the first off-treatment interval of intermittent androgen deprivation are prognostic for castration resistance in men with nonmetastatic prostate cancer. Clin Genitourin Cancer. 2015 Feb;13(1):10-6. doi: 10.1016/j.clgc.2014.08.003. Epub 2014 Aug 10. PMID 25242417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population for this trial was men with localized prostate cancer who had a rising PSA after definitive therapy (radiation therapy, brachytherapy, or radical prostatectomy). Patients were enrolled from Jan 1997 through Sept 2006 at the University of Washington and the Seattle Cancer Care Alliance.
Groups:
- Intermittent Androgen Suppression (IAS): Intermittent Androgen Suppression in 9 month cycles:
  1. Flutamide, 250 mg by mouth 3 times daily for a total of two weeks
  2. Leuprolide Acetate, 7.5mg intramuscular injections every 4 weeks for a total of nine months
Period: Overall Study
Arm/Group | Intermittent Androgen Suppression (IAS)
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intermittent Androgen Suppression (IAS): Intermittent Androgen Suppression in 9 month cycles with a combination of a two-week lead-in of Flutamide, followed by 9 monthly injections of Leuprolide Acetate.
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 102
Age, Continuous [Median (Full Range); unit: years] | 66 [60 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 98
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Time to Androgen Independence of Serum Prostate-Specific Antigen (PSA)
Description: Monthly Prostate-Specific Antigen (PSA) testing to assess the point at which each patient's disease stops responding to Androgen Deprivation Therapy (ADT). Androgen Independence (AI), also know as Castrate Resistance (CR), was defined as 2 serial rises in PSA while on ADT with Testosterone levels <50 ng/dL.
Time Frame: From date of first treatment until the date of development of CR, metastatic progression, or study withdrawal, whichever came first, assessed up to 16 years.
Population: 62 subjects were evaluable for this outcome measure, defined as having completed first cycle of ADT (9 months), having a measurable treatment break afterwards, and having sufficient PSA measurements to assess androgen independence.
Measure: Median (Full Range); unit: years
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 62
years | 4.0 [0.5 to 8.6]

2. Primary Outcome: Effect of IAS on Overall Survival.
Description: Assessment of overall survival measured as median time from completion of first full cycle of IAS until date of death from any cause.
Time Frame: From date of first treatment until the date of death or study withdrawal, whichever came first, assessed up to 16 years.
Population: 62 subjects were evaluable for this outcome measure, defined as having completed first cycle of ADT (9 months), having a measurable treatment break afterwards, and having sufficient data to assess survival status.
Measure: Median (Full Range); unit: years
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 62
years | 6.6 [2.9 to 13.0]

3. Secondary Outcome: Change in Standardized Bone Mineral Density (BMD) of the Spine During IAS
Description: Dual-energy x-ray absorptiometry (DEXA) scans were performed prior to first cycle of ADT, after completion of the first cycle of ADT, and prior to the start of the second cycle of ADT. Bone Mineral Density (BMD) was a assessed in g/cm^2 as a indicator of bone health for each patient at each time point.
Time Frame: From screening prior to first dose of ADT through the start of the second cycle of ADT.
Population: 56 subjects were evaluable for this outcome measure, defined as meeting all of the following: having completed first cycle of ADT (9 months); no prior or concurrent use of bisphosphonates; a minimum of 3 DEXA scans: prior to cycle 1, after cycle 1, and prior to cycle 2.
Measure: Number; unit: Percent change in BMD
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 56
Percent change in BMD
  Post Cycle 1 versus Baseline | -3.4
  Pre Cycle 2 versus Post Cycle 1 | 1.4

4. Secondary Outcome: Change in Standardized Bone Mineral Density (BMD) of the Left Hip During IAS
Description: Dual-energy x-ray absorptiometry (DEXA) scans were performed prior to first cycle of ADT, after completion of the first cycle of ADT, and prior to the start of the second cycle of ADT. Bone Mineral Density (BMD) was a assessed in g/cm^2 as a indicator of bone health. Percent change was assess for each patient at each time point.
Time Frame: From screening prior to first dose of ADT through the start of the second cycle of ADT.
Population: Out of 102 enrolled subjects, 56 were evaluable for this outcome measure, defined as having completed first cycle of ADT (9 months), no prior or concurrent use of bisphosphonates, and a minimum of 3 DEXA scans: prior to cycle 1, after cycle 1, and prior to cycle 2.
Measure: Number; unit: Percent change of BMD
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 56
Percent change of BMD
  Post Cycle 1 versus Baseline | -1.2
  Pre Cycle 2 versus Post Cycle 1 | -0.2

5. Secondary Outcome: Development of Osteopenia (Bone Loss) During IAS
Description: Dual-energy x-ray absorptiometry (DEXA) scans were performed prior to first cycle of ADT, after completion of the first cycle of ADT, and prior to the start of the second cycle of ADT. Bone Mineral Density (BMD) was a assessed in g/cm^2 as a indicator of bone health for each patient at each time point. This measure was defined as the percentage of participants with normal BMD scores at baseline who developed Osteopenia after the first cycle of ADT.
Time Frame: From screening prior to first dose of ADT through the start of the second cycle of ADT.
Population: 38 subjects were evaluable for this outcome measure, defined as meeting all of the following: having completed first cycle of ADT (9 months); no prior or concurrent use of bisphosphonates; a minimum of 3 DEXA scans: prior to cycle 1, after cycle 1, and prior to cycle 2; having baseline DEXA BMD within normal range at both spine and left hip.
Measure: Number; unit: percent of participants
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 38
percent of participants | 13.2

6. Secondary Outcome: Testosterone Levels During IAS
Description: Testosterone was measured at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: Sub-population of 20 evaluable patients, defined as having completed first cycle of ADT (9 months), having at least a 3 month treatment break afterwards, and having testosterone measurements at each of the listed time points.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
ng/ml
  Baseline | 406 (1.6)
  Measurement at Month 3 | 0.28 (0.24)
  Measurement at Month 9 | 0.20 (0.07)
  Measurement at Month 12 | 2.45 (1.35)

7. Secondary Outcome: Estradiol Levels During First Cycle of IAS
Description: Estradiol was measured at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: Sub-population of 20 evaluable patients, defined as having completed first cycle of ADT (9 months), having at least a 3 month treatment break afterwards, and having estradiol measurements at each of the listed time points.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
pg/ml
  Baseline | 33.60 (17.29)
  Measurement at Month 3 | 23.12 (6.56)
  Measurement at Month 9 | 22.76 (5.75)
  Measurement at Month 12 | 24.35 (6.46)

8. Secondary Outcome: Score on Spatial Ability Test (Block Design) During First Cycle of IAS
Description: Spatial Ability was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT. This assessment was based on the Wechsler Adult Intelligence Scale-Revised, Block Design sub-test and measures participants' ability to analyze and construct abstract figures from their component parts. The test allows a time limit of 3 minutes per design, for a total of nine designs. Score is based on total number of designs completed (max 9, min 0).
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: Sub-population of 20 evaluable patients, defined as having completed first cycle of ADT (9 months), having at least a 3 month treatment break afterwards, and having these neuro-psychological assessments at each of the listed time points.
Measure: Mean (Standard Deviation); unit: Number of correctly completed designs
Groups:
- Combined Androgen Blockade: Intermittent Hormone Therapy using Flutamide and Leuprolide acetate
  Flutamide: 250mg three times a day by mouth
  Leuprolide Acetate: 7.5mg once a month by intramuscular injection
Arm/Group | Combined Androgen Blockade
Number analyzed (Participants) | 20
Number of correctly completed designs
  Baseline | 8.65 (0.81)
  Score at Month 3 | 7.20 (1.21)
  Score at Month 9 | 8.82 (0.53)
  Score at Month 12 | 8.47 (1.06)

9. Secondary Outcome: Score on Spatial Ability Test (Mental Rotation) During First Cycle of IAS
Description: Spatial Ability (Mental Rotation) was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT. This assessment was based on the Vandenberg & Kuse (1978) Mental Rotation Test. Subjects are presented with line drawings of complex, three dimensional cubes on a computer screen. The subject must compare the two drawings and decide if they match. Score is based on number of correctly identified figures.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Number of correctly identified figures
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
Number of correctly identified figures
  Baseline | 16.12 (3.39)
  Score at Month 3 | 13.00 (3.01)
  Score at Month 9 | 16.52 (2.42)
  Score at Month 12 | 15.53 (3.08)

10. Secondary Outcome: Score on Executive Function Testing (Stroop Task) During First Cycle of IAS
Description: Executive Function was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT. This assessment was based on the Stroop Color Word Interference Task. Subjects are asked to read 100 color words (red, green, blue), followed by identification of color blocks followed by reading the color of the ink and ignoring the word (e.g., the word 'blue' printed in green letters). Assessment was based on the amount of time needed to time to complete the assessment.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: minutes to complete the assessment
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
minutes to complete the assessment
  Baseline | 51.00 (18.15)
  Score at Month 3 | 55.52 (22.11)
  Score at Month 9 | 47.58 (11.64)
  Score at Month 12 | 48.82 (13.31)

11. Secondary Outcome: Score on Verbal Memory Testing (Proactive Interference) During First Cycle of IAS
Description: Verbal Memory was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT via the Proactive Interference (PI) task. The PI task involves participants listening to a list of 10 words from the same semantic category (e.g., articles of clothing), and then recalling as many of these words as possible.The procedure is repeated for a total of 4 trials. Assessment is based on the total number of words recalled.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Number of correctly recalled words
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
Number of correctly recalled words
  Baseline | 21.31 (5.50)
  Score at Month 3 | 22.90 (5.03)
  Score at Month 9 | 22.70 (5.33)
  Score at Month 12 | 22.70 (4.33)

12. Secondary Outcome: Score on Visual Working Memory Test During First Cycle of IAS
Description: Visual Working Memory was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT. This task is based on the Subject Ordered Pointing Task (SOPT). The participant is shown a grid array of 10, 12 or 16 abstract designs and they must choose a new design with each refresh of the screen. Assessment is based on total number of errors.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: total number of errors
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
total number of errors
  Baseline | 13.22 (9.70)
  Score at Month 3 | 15.66 (8.50)
  Score at Month 9 | 12.35 (10.16)
  Score at Month 12 | 14.00 (11.04)

13. Secondary Outcome: Score on Verbal Memory Testing (Story Recall) During First Cycle of IAS
Description: Verbal Memory was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT via Story Recall. This task is based on the well known Wechsler Memory Scale -Revised Logical Memory task. Participants listened to two brief narratives (stories) and were asked to recall as much as possible immediately after hearing each story and following a 20-minute delay. Assessment was based on number of correctly recalled pieces of information after a delay.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: number of correctly recalled data points
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
number of correctly recalled data points
  Baseline | 35.06 (11.44)
  Score at Month 3 | 37.86 (12.11)
  Score at Month 9 | 39.38 (10.90)
  Score at Month 12 | 41.16 (8.08)

14. Secondary Outcome: Score on Spatial Memory Testing During First Cycle of IAS
Description: Spatial Memory was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT using the Puget Sound Route Learning Test. This test measured the ability to navigate a short route within a room. Three trials were administered followed by three trials of a new route using pictures placed on the floor as landmarks. A delayed recall is administered after twenty minutes. Performance was assessed based on number of correctly recalled sequences after a delay.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: number of correctly recalled sequences
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
number of correctly recalled sequences
  Baseline | 19.50 (10.05)
  Score at Month 3 | 22.00 (9.39)
  Score at Month 9 | 23.76 (8.60)
  Score at Month 12 | 24.12 (8.86)

15. Secondary Outcome: Score on Verbal Ability/Fluency Testing During First Cycle of IAS
Description: Verbal Ability/Fluency was assessed at baseline, and at Month 3, Month 9, and Month 12 after the start of the first cycle of ADT. Participants were asked to verbally generate as many words beginning with a particular letter (e.g. P) within a 60 second period. Two trials were administered with two different letters. The total number of words generated was recorded for each letter and summed and analyzed.
Time Frame: Baseline, Month 3, Month 9, and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Number of words generated
Arm/Group | Intermittent Androgen Suppression (IAS)
Number analyzed (Participants) | 20
Number of words generated
  Baseline | 24.65 (7.11)
  Score at Month 3 | 26.15 (9.14)
  Score at Month 9 | 26.29 (7.44)
  Score at Month 12 | 25.70 (8.29)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for each patient from the start of treatment until discontinuation from the study, an average of 16 years per patient.
Arm/Group | Combined Androgen Blockade
All-Cause Mortality (participants affected / at risk) | 33/102
Serious Adverse Events (participants affected / at risk) | 5/102
Other Adverse Events (participants affected / at risk) | 91/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Androgen Blockade (N=102)
pnemonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 1 (3)
Atrioventricular node ablation (Cardiac disorders) | 1 (1)
exacerbation of claudication (Musculoskeletal and connective tissue disorders) | 1 (1)
stroke (Nervous system disorders) | 1 (1)
left hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Androgen Blockade (N=102)
depression (Psychiatric disorders) | 5 (102)
fatigue (General disorders) | 9 (102)
hot flashes (General disorders) | 14 (102)
hyperlipidemia (Investigations) | 9 (102)
hypertension (Cardiac disorders) | 6 (102)
urinary incontinence (Renal and urinary disorders) | 12 (102)
nocturia (Renal and urinary disorders) | 15 (102)
osteopenia (Musculoskeletal and connective tissue disorders) | 5 (102)
pain, bone and muscle (Musculoskeletal and connective tissue disorders) | 6 (102)
renal insufficiency (Renal and urinary disorders) | 5 (102)
weight gain (General disorders) | 6 (102)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No